CLINICAL TRIAL: NCT04790513
Title: Randomized, Open-label, Phase 3 Study to Evaluate the Efficacy and Safety of LIB003, Evolocumab and Alirocumab in CVD Patients, or at High Risk for CVD, on Stable Lipid-Lowering Therapy Requiring Additional LDL-C Reduction (LIBerate-H2H)
Brief Title: Trial to Evaluate Efficacy and Safety of LIB003, Evolocumab and Alirocumab in High-risk CVD Patients
Acronym: LIBerate-H2H
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIB003-011
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Hypercholesterolemia; Cardiovascular Diseases
Keywords: lerodalcibep; evolocumab; alirocumab
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — evolocumab; alirocumab

STUDY DESIGN:
Intervention Model Description: randomized, open-label with blinded lipid levels
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: lipid levels measured and central laboratory will be blinded to participants, investigators, and sponsor, DSMB and CEC (Cardiovascular Events Committee)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LIB003 (lerodalcibep) (Experimental): 300 mg SC Q4W
  Interventions: Biological: lerodalcibep
- evolocumab (Active Comparator): 420 mg SC Q4W
  Interventions: Biological: evolocumab
- alirocumab (Active Comparator): 300 mg SC Q4W
  Interventions: Biological: alirocumab

INTERVENTIONS:
Biological: lerodalcibep — anti-PCSK9 small binding protein
  Other Names: LIB003
  Arms: LIB003 (lerodalcibep)
Biological: evolocumab — monoclonal antibody to PCSK9
  Other Names: Repatha
  Arms: evolocumab
Biological: alirocumab — monoclonal antibody to PCSK9
  Other Names: Praluent
  Arms: alirocumab

SUMMARY:
Comparison of LDL-C reductions at Week 12 of monthly (Q4W[≤ 31 days]) dosing of LIB003 300 mg administered subcutaneously (SC) to Q4W dosing of evolocumab (Repatha) 420 mg and alirocumab (Praluent) 300 mg in patients with CVD or at high risk for CVD on a stable diet and high intensity statin and other LDL-C-lowering drug therapy.

DETAILED DESCRIPTION:
This is a randomized, open-label Phase 3 study of 12 weeks duration comparing Q4W SC doses of LIB003 300 mg, evolocumab (Repatha) 420 mg and alirocumab (Praluent) 300 mg. Approximately 220 males and females aged ≥18 years who fulfill all of the inclusion and exclusion criteria will be enrolled at up to 25 sites in the United States. Patients will be stratified by baseline LDL-C and randomized in a 2:2:1 ratio to LIB003 (88 patients), Repatha (88 patients) or Praluent (44 patients) administered SC Q4W (≤31 days). The study will consist of a Screening Period and a Treatment Period. The total study duration will be up to 21 weeks which includes up to 9-week Screening Period (depending on period required for washout of PCSK9 mAb and/or intensification of statin treatment) and 12 weeks of study drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* diagnosed with CVD or a high risk of CVD based on 2019 ESC/EAS guidelines
* Weight of ≥40 kg (88 lb) and body mass index (BMI) ≥17 and ≤42 kg/m2
* LDL-C ≥90 mg/dL and TG ≤400 mg/dL while on stable diet & lipid-lowering oral drug therapy (ie, high intensity statin with or without ezetimibe) and no PCSK9 mAb for 4 weeks if previously on Q2W dosing or 8 weeks if on Q4W dosing.
* Females of childbearing potential must be using a highly effective form of birth control if sexually active and have a negative urine pregnancy test at the last Screening Visit

Exclusion Criteria:

* at screening visit: not on high intensity statin; mipomersen or lomitapide within 6 months; gemfibrozil within 6 weeks; bempedoic acid within 4 weeks; inclisiran within 12 months; apheresis within 8 weeks
* HoFH defined clinically and/or genetically
* History of prior or active clinical condition or acute and/or unstable systemic disease compromising patient inclusion, at the discretion of the Investigator
* estimated glomerular filtration rate <30 mL/min/1.73m2 at screening
* Active liver disease or hepatic dysfunction, history of liver transplant, and/or AST or ALT >2.5 × the ULN
* Uncontrolled Type 1 or Type 2 diabetes mellitus, defined as fasting glucose ≥200 mg/dL or glycated hemoglobin (HbA1c) of ≥9%
* NY Heart Association class III-IV heart failure; or patients with last documented left ventricular ejection fraction <30%; planned PCI, CABG or cardiac surgery
* Uncontrolled hypertension defined as evidenced by a reproducible (repeated 5 minutes apart) sitting blood pressure ≥160 mmHg systolic or ≥100 mmHg diastolic;
* Enrolled in another investigational device or drug study, or less than 30 days or 5 half-lives since ending another investigational device or drug study(ies), or receiving PCSK9 or Lp(a) siRNA or locked nucleic acid-reducing agents within 12 months of the Screening Visit;
* Have any other finding which, in the opinion of the Investigator, would compromise the patient's safety or participation in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
LDL-C reduction from baseline at 12 weeks | 12 weeks
  LS Mean percent change from baseline to week 12

SECONDARY OUTCOMES:
Achieved ESC/EAS LDL-C goals | 12 weeks
  Percent of patients achieving ESC/EAS 2019 LDL-C target
tolerability and safety of each treatment: injection site reactions | 12 weeks
  ISR (injection site reactions) after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Evan A Stein, MD PhD, Study Director — LIB Therapeutics
Locations (3):
- United States (3):
  - Sterling Research Group, Cincinnati, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Metabolic & Atherosclerosis Research Center (MARC), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No